CLINICAL TRIAL: NCT02356042
Title: Effects of Geriatric Inclusive Art Activity in Nursing Home Residents (GIA)
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Cémavie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013-42
Record Dates: First submitted 2015-01-26; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-01

CONDITIONS: Geriatric Disorders
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Nursing home residents practicing GIA activity
  Interventions: Other: Geriatric inclusive art (GIA) activity
- Nursing home residents no practicing GIA activity

INTERVENTIONS:
Other: Geriatric inclusive art (GIA) activity — The frequency of GIA sessions in this study was from 1 to 2 per month. The time of a session was around 1 hour 30 minutes. Participants of intervention group benefited GIA activity during a 6-month follow-up period.
  Groups: Nursing home residents practicing GIA activity

SUMMARY:
The study aimed to compare the changes in health and functional status between nursing home residents practicing GIA activity and a control group of residents, and to examine the changes in residents' abilities to participate in GIA activity.

DETAILED DESCRIPTION:
Geriatric inclusive art (GIA) activity is a derived form of art therapy using painting to make older adults aware of their abilities through an improvement of emotional well-being (1). GIA protected against in-hospital mortality in demented older inpatients and has also been associated with shorter length of hospital stay in geriatric inpatients. These GIA-related positive effects suggest that GIA activity may improve health and functional status in the elderly. To date, effects of GIA on health and functional status in nursing home residents have not been examined.

Based on the previous positive effects reported in older inpatients practicing GIA activity, the investigators hypothesized that GIA activity could improve health and/or functional status of nursing homes residents.

ELIGIBILITY:
Inclusion Criteria:

* Being a resident in the nursing home "la Grande Providence" (Nantes - Loire Atlantique, France)
* Ability to answer questions
* Being affiliated to the French health insurance

Exclusion Criteria:

* Inability to understand and speak French
* Opposition to the use of information collected for research purposes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were recruited in nursing home.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in health and functional status measured by a standardized questionnaire | This outcome is assessed at baseline and at 6 months
  Change in health and functional status was measured by a standardized questionnaire

SECONDARY OUTCOMES:
Change in the number of drugs daily taken assessed by a standardized questionnaire | This outcome is assessed at baseline and at 6 months
  The number of drugs daily taken was assessed by a standardized questionnaire
History of falls in the past 6 months assessed by a standardized questionnaire | This outcome is assessed at baseline and at 6 months
  History of falls was assessed by a standardized questionnaire
Have an unscheduled medical consultation assessed by a standardized questionnaire | This outcome is assessed at baseline and at 6 months
  Unscheduled medical consultation was assessed by a standardized questionnaire
Being hospitalized unscheduled manner assessed by a standardized questionnaire | This outcome is assessed at baseline and at 6 months
  Unscheduled hospitalization was assessed by a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Fondation Cémavie, Nantes, France